CLINICAL TRIAL: NCT04296565
Title: Water-based Activity to Enhance Recall in Veterans: A Randomized Clinical Trial
Brief Title: Water-based Activity to Enhance Recall in Veterans
Acronym: WATER-Vet
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E3143-R; 1I01RX003143-01A2 (NIH)
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Cognition; Alzheimer's Disease; Physical Exercise; Cognitive Training
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Other): Usual Care condition involves receipt of educational materials about brain health and healthy lifestyles as well as regular contact with study staff.
  Interventions: Behavioral: Usual Care
- WATER+CT (Experimental): This is an 8 month long two phase intervention. The first phase consists of 6 months of thrice weekly pool based physical activity occurring at the Palo Alto VA Health Care System. After completion of the 6 month long water based physical activity, participants transition to a ten session cognitive training program at the Palo Alto VA. The cognitive training classes are approximately two hours in length and will be spread over ten sessions across 4 weeks.
  Interventions: Behavioral: WATER+CT

INTERVENTIONS:
Behavioral: Usual Care — Usual Care condition involves receipt of educational materials about brain health and healthy lifestyles as well as regular contact with study staff
  Arms: Usual Care
Behavioral: WATER+CT — This is an 8 month long two phase intervention. The first phase consists of 6 months of thrice weekly pool based physical activity occurring at the Palo Alto VA Health Care System. After completion of the 6 month long water based physical activity, participants transition to a ten session cognitive training program at the Palo Alto VA. The cognitive training classes are approximately two hours in length and will be spread over ten sessions across 4 weeks.
  Arms: WATER+CT

SUMMARY:
This four-year study will evaluate the efficacy of an exercise training augmentation for cognitive training intervention to improve memory performance in Veterans with a diagnosis of amnestic Mild Cognitive Impairment (aMCI). This is a two-phased trial: 1) an exercise phase and 2) a cognitive training program. The exercise phase will be an aquatic based exercise program. A combination of exercise and cognitive training programs designed for persons without cognitive impairment have significantly improved memory more than other single intervention groups (exercise only, cognitive training only) and given the success of combination training programs with healthy older adults, it is important to adapt these programs for persons beginning to exhibit clinically significant memory problems, such as those with aMCI.

DETAILED DESCRIPTION:
The primary research question of the proposed study is this: Is a water-based exercise plus cognitive training intervention efficacious in improving cognitive outcomes for Veterans with Mild Cognitive Impairment (MCI)? The investigators address the need to improve cognitive function in this vulnerable population through a novel multi-component training program that will combine two interventions: water-based exercise and cognitive training. The proposed four-year randomized controlled trial will compare water-based exercise + cognitive training (WATER+CT) to a Usual Care Control Condition (UC). The primary aim of the proposed research is to evaluate the efficacy of WATER+CT to improve cognitive function in Veterans with MCI. Secondary aims of the proposed research are: 1) to evaluate the efficacy of WATER+CT to improve peak oxygen consumption and 2) to evaluate the durability of the cognitive benefits derived from WATER+CT. Exploratory aims of the proposed research are to evaluate moderators and mediators of treatment response.

These aims will be tested in a single-blind randomized controlled trial that will compare the efficacy of WATER+CT to UC. This trial will include 130 Veterans meeting criteria for MCI age 50-90 with half randomized to WATER+CT and half randomized to UC. For the WATER+CT condition, the exercise training (i.e., WATER) consists of a six-month long individualized exercise program of water-based exercises. During this phase, Veterans will come to thrice-weekly group sessions at Aquatic Therapy Center at the VA Palo Alto Health Care System (VAPAHCS). After completion of the exercise program, Veterans will begin classroom-based cognitive training at the VAPAHCS for up to two months. The CT is based on an efficacious training program that is structured around two components, pre-training and mnemonic training, both of which have been used successfully in persons with MCI. Veterans randomized to the UC control condition will receive educational materials about brain health in addition to their usual care, which is the care they would typically receive in the VA. After completion of the active treatment phase, Veterans will transition to the six-month long follow-up phase. At the end of the six-month long follow-up phase, participants will return to the VA for a final follow-up visit.

Participants will complete a variety of neuropsychological measures taping into areas of cognition such as attention, executive functioning, and memory. Participants will also undergo physical fitness assessments including a 6-minute walk test and an exercise treadmill test. To study possible predictors of response to treatment, the investigators will also collect biological (cardiovascular functioning and BDNF plasma levels) and genetic data (APOE and BDNF genotypes) from these participants. The investigators hope to provide evidence of the efficacy of an exercise training augmentation for cognitive training thus laying the groundwork for future VA health care system wide deployment of a lifestyle intervention to prevent Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Veterans, aged 50 to 90, of any racial or ethnic group
* Diagnosis of single or multi-domain amnestic MCI using criteria per National Institute on Aging/Alzheimer's Association Guidelines
* Available informant for completion of the Clinical Dementia Rating Scale
* Visual and auditory acuity to allow neuropsychological testing
* Willingness to participate in clinical trial for 14 months (8-month treatment phase, 6-month no-contact follow-up phase)
* Musculoskeletal illness or injury (i.e., osteoporosis, degenerative disc or joint disease, arthritis, obesity)
* Approval by Primary Care Provider to participate in water-based physical exercise

Exclusion Criteria:

Psychiatric Exclusions

* Current, uncontrolled severe psychiatric disorder, such as Bipolar I, Schizophrenia, or Major Depressive Disorder as determined by the Mini International Neuropsychiatric Interview (MINI)
* Diagnosis of dementia, Clinical Dementia Rating Scale (CDR) > 0.5; modified Hachinksi score 4; or delirium. Those Veterans with scores indicative of dementia (CDR > 0.5, modified Hachinksi 4) will be referred to the Memory Disorders Clinic at VAPAHCS for a full diagnostic work-up

Medical Exclusions

* History of neurological (e.g., multiple sclerosis, seizure disorder, stroke,) or system illness affecting CNS function (e.g., liver failure, kidney failure, congestive heart failure, systemic cancer)
* Acute illness or unstable chronic illness, e.g., history of severe liver disease (cirrhosis, esophageal varices, ascites, portal hypertension, hepatic encephalopathy)
* Current severe cardiac disease (e.g., uncontrolled atrial fibrillation, defined as mean 24 hour heart rate >85 beats/min, or 24 hour maximal ventricular rate >150 beats/min; uncontrolled ventricular arrhythmias, defined as recurrent ventricular tachycardia >3 beats in succession, or 24 hour PVC count >20%; active pericarditis or myocarditis; Class III/IV heart failure and / or ejection fraction < 20%; thrombophlebitis; pulmonary disease with a drop in O2 Sat with exercise to 90% without oxygen; embolism within past 6 months)
* Inability to participate in an exercise stress test
* Inability to read, verbalize understanding and voluntarily sign the Informed Consent

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function Composite Score (ADAS-Cog-Exe) | 8 months
  The ADAS-Cog is a structured scale that evaluates multiple cognitive domains including: orientation, memory, reasoning, language, and praxis.

SECONDARY OUTCOMES:
Peak VO2 | 8 months
  Peak VO2, or VO2Max, is defined as the minute volume of O2 utilization

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kaci Fairchild, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No